CLINICAL TRIAL: NCT06085417
Title: Comparison of the Effects of Dexamethasone and magnesıum Sulphate Used as Adjuvant in Infraclavicular Brachial Plexus Nerve Block.
Brief Title: Comparison of the Effects of Dexamethasone and magnesıum Sulphate Used as Adjuvant in Infraclavicular Nerve Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacı Yusuf Güneş, MD, Assistant proffesor, Yuzuncu Yil University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 03.03.2022/03
Record Dates: First submitted 2023-09-19; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Bupivacaine; Dexamethasone; Magnesıum Sulphate; Adjuvant
Keywords: Adjuvant; Bupivacaine; Dexamethasone; Infraclavicular brachial plexus nerve block; Magnesıum sulphate
MeSH Terms: interventions — Bupivacaine; Dexamethasone; blood-group-substance alpha-D-galactosyltransferase; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: The required asepsis in the area where the block would be applied was provided with 10% poviodine iodine and covered with a sterile drape. The USG probe was placed in the sagittal plane 1 cm below the intersection point between the coracoid process and the clavicle, and after visualizing the lateral, posterior and medial cords around the axillary artery, a peripheral nerve block needle was directed towards the 8 o'clock position relative to the axillary artery, in the same plane as the USG probe. When the expected distal motor response was obtained, the current of the peripheral nerve stimulator was reduced to 0.3 mA to avoid intraneural injection. If the motor response disappeared, local anesthetic was injected slowly. Sensory and motor block onset times, saturation, systolic blood pressure, diastolic blood pressure, mean arterial pressure and heart rate peak values at the 0th, 15th, 30th and 60th minutes after the block were recorded.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group B (bupivacaine) (n= 30) (Sham Comparator): For Group B (control group), 100 mg bupivacaine hydrochloride+ isotonic saline (5ml) was administered in a total volume of 25 ml. Patients' ASA score, demographic data (age, height, weight), systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, SpO₂, sensory and motor block onset times , need for additional sedation, side effects and complications, if any, were recorded. The patients' postoperative sensory block and motor block resolution times, VAS scores at the 0th, 3rd, 6th, 12th and 24th postoperative hours, total opioid and NSAID requirements in the first 24 hours, and analgesia durations were recorded.
  During the perioperative period, all patients were monitored for side effects such as nausea, vomiting, tinnitus, metallic taste in the mouth, and drug allergy.
  Interventions: Drug: bupivacaine
- Group Group B+D (bupivacaine + dexamethasone group) (n= 30) (Experimental): For Group B+D (bupivacaine + dexamethasone group), 100 mg bupivacaine hydrochloride + 4 mg dexamethasone phosphate+ isotonic saline (4 ml) was administered in a total volume of 25 ml. Patients' ASA score, demographic data (age, height, weight), systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, SpO₂, sensory and motor block onset times , need for additional sedation, side effects and complications, if any, were recorded. The patients' postoperative sensory block and motor block resolution times, VAS scores at the 0th, 3rd, 6th, 12th and 24th postoperative hours, total opioid and NSAID requirements in the first 24 hours, and analgesia durations were recorded. During the perioperative period, all patients were monitored for side effects such as nausea, vomiting, tinnitus, metallic taste in the mouth, and drug allergy.
  Interventions: Drug: Bupivacaine + dexamethasone
- Group B+M (bupivacaine + magnesium group) (n= 30) (Active Comparator): For Group B+M (bupivacaine + magnesium group), 100 mg bupivacaine hydrochloride (20ml 0.5% marcaine aspen, turkey) + 150 mg magnesium sulfate (1ml 15% magnesium sulfate, onfarma, turkey) + isotonic saline (4 ml) was administered in a total volume of 25 ml. Patients' ASA score, demographic data (age, height, weight), systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, SpO₂, sensory and motor block onset times , need for additional sedation, side effects and complications, if any, were recorded. The patients' postoperative sensory block and motor block resolution times, VAS scores at the 0th, 3rd, 6th, 12th and 24th postoperative hours, total opioid and NSAID requirements in the first 24 hours, and analgesia durations were recorded.
  During the perioperative period, all patients were monitored for side effects such as nausea, vomiting, tinnitus, metallic taste in the mouth, and drug allergy.
  Interventions: Drug: Bupivacaine + magnesium sulphate

INTERVENTIONS:
Drug: Bupivacaine + dexamethasone — Vital signs were recorded before the block. Peripheral vascular access was established with a 20-gauge catheter and 0.9% NaCl crystalloid solution infusion was started. For sedation, all patients were routinely administered 1mg midazolam intravenously before the procedure. Patients' ASA score, demographic data (age, height, weight), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), SpO₂, sensory and motor block onset times , need for additional sedation, side effects and complications, if any, were recorded. The patients' postoperative sensory block and motor block resolution times, VAS scores at the 0th, 3rd, 6th, 12th and 24th postoperative hours, total opioid and NSAID requirements in the first 24 hours, and analgesia durations were recorded.
  During the perioperative period, all patients were monitored for side effects such as nausea, vomiting, tinnitus, metallic taste in the mouth, and drug allergy.
  Other Names: Group B+D
  Arms: Group Group B+D (bupivacaine + dexamethasone group) (n= 30)
Drug: Bupivacaine + magnesium sulphate — Vital signs were recorded before the block. Peripheral vascular access was established with a 20-gauge catheter and 0.9% NaCl crystalloid solution infusion was started. For sedation, all patients were routinely administered 1mg midazolam intravenously before the procedure. Patients' ASA score, demographic data (age, height, weight), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), SpO₂, sensory and motor block onset times , need for additional sedation, side effects and complications, if any, were recorded. The patients' postoperative sensory block and motor block resolution times, VAS scores at the 0th, 3rd, 6th, 12th and 24th postoperative hours, total opioid and NSAID requirements in the first 24 hours, and analgesia durations were recorded.
  During the perioperative period, all patients were monitored for side effects such as nausea, vomiting, tinnitus, metallic taste in the mouth, and drug allergy.
  Other Names: Group B+M
  Arms: Group B+M (bupivacaine + magnesium group) (n= 30)
Drug: bupivacaine — bupivacaine
  Arms: Group B (bupivacaine) (n= 30)

SUMMARY:
The aim of this prospective clinical study is to compare the effectiveness of dexamethasone and magnesium sulfate added as adjuvants to bupivacaine in infraclavicular brachial plexus block used under ultrasound guidance for upper extremity surgeries.

DETAILED DESCRIPTION:
This study was conducted on 90 patients who underwent upper extremity surgery under infraclavicular brachial plexus block.

90 patients included in the study were randomized into 3 groups of 30 people each by the sealed envelope method.

30 participants were included in Group Bupivacaine, 30 participants were included in Group Bupivacaine + Dexamethasone and 30 participants were included in Group Bupivacaine + Magnesium sulfate.

The study was started as double blind. According to the local anesthetic used, patients were group B (30 patients, 20 cc 0.5% bupivacaine + 5 cc 0.9% NaCl), group B+D (30 patients, 20 cc 0.5% bupivacaine + 4 mg dexamethasone + 4 cc 0.9% NaCl), group They were divided into three groups as B+M (30 patients, 20 cc 0.5% bupivacaine + 150 mg magnesium sulfate + 4 cc 0.9% NaCl).

Complications of the patients, such as sensory block and motor block onset times, peroperative hemodynamic parameters, need for additional analgesia, postoperative block duration, analgesia duration, opioid and NSAID consumption, nausea and vomiting, were recorded

ELIGIBILITY:
Inclusion Criteria:

* Participants providing informed written and verbal consent
* 18-65 years old
* ASA I-II
* Cases undergoing elective upper extremity surger

Exclusion Criteria:

* Cases that do not accept regional anesthesia application
* Those who are under 18 years of age and over 65 years of age
* ASA III and above
* Cases in which the operation was started with infraclavicular block and then transferred to general anesthesia.
* Those with liver and kidney dysfunction
* Those with diabetes mellitus
* Those with drug allergies
* Patients with acid-base and electrolyte disorders
* Pregnant women
* Emergency cases
* Those with neuropathic disorders
* Those with significant psychiatric and cognitive disorders or substance addiction
* Those with a history of clavicle fracture, pneumonectomy, contralateral hemidiaphragmatic paralysis, pneumothorax, phrenic or recurrent laryngeal nerve palsy.
* Cases with BMI>30 or BMI<18
* Patients in whom regional anesthesia was contraindicated (sepsis, local infection, coagulopathy, heart disease, hypovolemia) were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Motor block onset time | 24 hours
  Motor block examination was performed with the modified Bromage scale. In the motor block examination, thumb orientation was examined for the median nerve, thumb abduction for the radial nerve, thumb adduction for the ulnar nerve, and elbow flexion for the musculocutaneous nerve. Patients with a modified Bromage scale ≤ 2 on the side where the block was applied were considered to have a successful block and the patient's surgery was initiated.
Motor Block Duration | 24 hours
  Motor block durations were determined according to the Bromage scales at the 1st, 3rd, 6th, 12th and 24th postoperative hours.
Sensory block onset time | 24 hours
  Pinprick sensory test was used in the sensory examination of the patients. Sensory examination was performed using a pinprick test on the first 3 fingers and the dorsal side of the wrist for the radial nerve, the medial side of the 5th finger for the ulnar nerve, the first 3 fingers and the volar side of the wrist for the median nerve, and the lateral region of the forearm for the musculocutaneous nerve.Pinprick sensory test ≤ 1 on the side where the block was applied were considered to have a successful block and the patient's surgery was initiated.
Sensory block duration | 24 hours
  Sensory block durations were determined according to the Pinprick sensory test at the 1st, 3rd, 6th, 12th and 24th postoperative hours.
VAS score | 24 hours
  VAS scores at the 1st, 3rd, 6th, 12th and 24th postoperative hours were evaluated. Dexketoprofen trometamol 50 mg was given intravenously to patients with a postoperative VAS Score of 4 and above. If the VAS Score was 6 or above even though NSAIDs were administered, the patients were given the opioid analgesic tramadol hydrochloride 1 mg/kg intravenously.

CONTACTS AND LOCATIONS:
Overall Officials: Haci Y GUNES, Assist.prof, Principal Investigator — Van Yüzüncü Yıl University Van, Turkey
Locations (1):
- Haci Yusuf GUNES, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be share for other resarchers.
Supporting Information: Study Protocol, SAP
Time Frame: 6 month
Access Criteria: The access can be provided via the e-mail addresses below hyusufgunes@hotmail.com

REFERENCES:
- [Background] Mirza F, Brown AR. Ultrasound-guided regional anesthesia for procedures of the upper extremity. Anesthesiol Res Pract. 2011;2011:579824. doi: 10.1155/2011/579824. Epub 2011 May 30. PMID 21716734
- [Background] O'Donnell BD, Ryan H, O'Sullivan O, Iohom G. Ultrasound-guided axillary brachial plexus block with 20 milliliters local anesthetic mixture versus general anesthesia for upper limb trauma surgery: an observer-blinded, prospective, randomized, controlled trial. Anesth Analg. 2009 Jul;109(1):279-83. doi: 10.1213/ane.0b013e3181a3e721. PMID 19535722
- [Background] Klaastad O, Sauter AR, Dodgson MS. Brachial plexus block with or without ultrasound guidance. Curr Opin Anaesthesiol. 2009 Oct;22(5):655-60. doi: 10.1097/ACO.0b013e32832eb7d3. PMID 19550303